CLINICAL TRIAL: NCT07403786
Title: Urethral Resistive Index (URI): A New Uroflowmetric Parameter in the Non-Invasive Diagnosis of Urethral Obstruction
Brief Title: Urethral Resistive Index (URI): A New Parameter for Diagnosing Urethral Obstruction
Acronym: URI
Status: Not yet recruiting | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Yusuf Gökkurt, Attending Physician, Department of Urology, Ankara City Hospital Bilkent
Other Study IDs: TABED 1/2090/2026
Record Dates: First submitted 2026-02-05; First posted 2026-02-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Urethral Stricture
MeSH Terms: conditions — Urethral Stricture

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Stricture Group: Patients with suspected urethral stricture scheduled for surgery (urethroplasty or internal urethrotomy), with the diagnosis confirmed intraoperatively.
  Interventions: Diagnostic Test: Uroflowmetry with URI Calculation
- Control Group: Healthy male volunteers in a similar age range as the stricture group, without any lower urinary tract symptoms.
  Interventions: Diagnostic Test: Uroflowmetry with URI Calculation

INTERVENTIONS:
Diagnostic Test: Uroflowmetry with URI Calculation — Performing natural and forced (Valsalva) uroflowmetry sessions to calculate the Urethral Resistive Index.

SUMMARY:
This prospective observational study aims to evaluate the diagnostic accuracy of a new, non-invasive uroflowmetry parameter called the Urethral Resistive Index (URI) for detecting urethral stricture in men. Currently, diagnosing urethral stricture often requires invasive procedures like surgery or pressure-flow studies. This research seeks to develop URI as a practical and painless screening tool that could reduce the need for such invasive interventions.

Study Procedures:

A total of 60 male participants (30 with suspected urethral stricture and 30 healthy volunteers) will be enrolled. Participants will undergo two standard, non-invasive uroflowmetry (voiding) tests. The first test is a routine natural voiding session. The second test involves a "forced voiding" (Valsalva maneuver) once the participant feels a sufficient urge to urinate again. The URI is then calculated by comparing the flow rates of these two sessions.

Goals and Benefits: The primary goal is to determine the optimal "cut-off" value of the URI that accurately identifies a surgically proven urethral stricture. By demonstrating URI's effectiveness, the study aims to expedite the diagnostic process and spare patients from unnecessary invasive tests. The procedure involves minimal risk, primarily temporary discomfort or psychological stress during the voiding tests

DETAILED DESCRIPTION:
This methodological study is designed as a prospective, cross-sectional, and observational diagnostic accuracy study. The primary objective is to evaluate the clinical validity of the Urethral Resistive Index (URI), a novel non-invasive parameter, in the diagnosis of urethral stricture.

Study Population and Groups:

The study will include a total of 60 male participants aged between 18 and 80 years.

Stricture Group (n=30): Patients planned for surgery (urethroplasty or internal urethrotomy) due to suspected urethral stricture, where the presence of the stricture is confirmed intraoperatively.

Control Group (n=30): Healthy male volunteers without lower urinary tract symptoms, matched for age.

Methodology: The study focuses on comparing standard uroflowmetry with "forced" uroflowmetry using the Valsalva maneuver. All clinical and uroflowmetric parameters will be collected at the Ankara Bilkent City Hospital Urology Clinic.

Natural Uroflowmetry: Participants will perform a standard uroflowmetry test. Forced Uroflowmetry: After reaching sufficient bladder fullness again, participants will perform a second test using the Valsalva maneuver (forced voiding).

Calculation: The URI will be calculated using the formula:

URI= Qmax,forced/ Qmax,normal

Statistical Analysis: The diagnostic performance of the URI will be evaluated using Receiver Operating Characteristic (ROC) curve analysis. The Area Under the Curve (AUC) will be calculated, and the optimal cut-off value for determining urethral stricture will be identified with corresponding sensitivity and specificity values. Correlation between URI and clinical symptom scores, such as the International Prostate Symptom Score (IPSS), will also be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Male participants aged between 18 and 80 years.
* For the Stricture Group: Patients scheduled for surgery (urethroplasty or internal urethrotomy) due to suspected urethral stricture, where the diagnosis is confirmed intraoperatively.
* For the Control Group: Healthy male volunteers without any lower urinary tract symptoms.
* Voluntary signing of the Informed Consent Form.

Exclusion Criteria:

* Voiding volume less than 150 mL.
* Causes of obstruction other than stricture, such as Benign Prostatic Hyperplasia (BPH).
* Diagnosis of neurogenic bladder dysfunction or a history of neurological disease affecting bladder function.
* Presence of severe comorbidities.

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population consists of 60 male participants, aged 18 to 80 years, recruited from the Urology Outpatient Clinic at Ankara Bilkent City Hospital. The population is divided into two distinct groups: a Stricture Group (n=30) comprising patients with suspected urethral stricture whose diagnosis is confirmed intraoperatively during scheduled surgery, and a Control Group (n=30) comprising healthy male volunteers with a similar age distribution and no lower urinary tract symptoms. Participants are selected based on their clinical presentation and willingness to undergo a specialized two-stage uroflowmetry protocol.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2026-02-09 (Estimated); Primary Completion 2026-05-10 (Estimated); Study Completion 2026-07-10 (Estimated)

PRIMARY OUTCOMES:
Urethral Resistive Index (URI) | At the time of the uroflowmetry procedure (Baseline)
  A novel non-invasive uroflowmetric parameter calculated to assess the resistance of the urethra during voiding. It is derived using the formula: URI=Qmax,natural/Qmax,forced.

IPD SHARING:
Plan to Share IPD: No
To protect participant privacy and maintain data confidentiality according to local institutional regulations

REFERENCES:
- [Background] Kranse R, van Mastrigt R. Bladder outlet resistance. J Urol. 2003 Mar;169(3):1007-10. doi: 10.1097/01.ju.0000052693.58772.23. PMID 12576832
- [Background] Spyropoulos E, Galanakis I, Deligiannis D, Spyropoulou A, Kotsiris D, Panagopoulos A, Mavrikos S. Flow resistive forces index (QRF): Development and clinical applicability assessment of a novel measure of bladder outlet resistance, aiming to enhance the diagnostic performance of uroflowmetry. Low Urin Tract Symptoms. 2020 Sep;12(3):190-197. doi: 10.1111/luts.12301. Epub 2020 Jan 30. PMID 31999073
- [Background] Krukowski J, Kaluzny A, Klacz J, Piatkowska A, Matuszewski M. Evaluation of non-invasive tests as diagnostic tools in assessment of bladder outlet obstruction severity in men with anterior urethral stricture. Cent European J Urol. 2021;74(3):422-428. doi: 10.5173/ceju.2021.3.153.R1. Epub 2021 Jul 27. PMID 34729232